CLINICAL TRIAL: NCT00429013
Title: A Prospective, Randomised, Controlled, Open Study. Phase II Treatment Equivalent.
Brief Title: Pressure Ulcer Formation Prevention in Paraplegics Using Computer and Sensory Substitution Via the Tongue.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: principal criteria was achieved with the intermediate statistical analysis
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Centre Medico Universitaire Daniel Douady (CMUDD) (Other); TIMC-IMAG (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DCIC-05-44
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: PARAPLEGIA
Keywords: Pressure ulcer; Lingual electric stimulation; Paraplegic patient; Pressure Ulcer/Prevention & control
MeSH Terms: conditions — Paraplegia; Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (No Intervention): no medical device
- 1 (Experimental): medical device
  Interventions: Device: Tongue Display Unit

INTERVENTIONS:
Device: Tongue Display Unit — lingual electric stimulation
  Arms: 1

SUMMARY:
Will the use of sensory substitution by lingual electric stimulation improve in a suitable way, for paraplegic subject, the spatial distribution of pressure applied at the seat/skin interface in order to prevent the formation of pressure ulcer? We will try to demonstrate that paraplegic subject move in an appropriate matter, in term of pressure, after a movement way advised by periodical electric stimuli on the tongue.

DETAILED DESCRIPTION:
The objective of this study will be, to validate or not, the possibility to inform, in a suitable way, paraplegic subject by a lingual electric stimulation.

Two A and B study groups of paraplegic subjects will be built-up in a randomized way. Under standardized conditions, the A study group subject will modify his usual behavior by using the cosmetically acceptable interface to get back information for moving his chest in a suitable way in order to correct identified maxima of pressure at the seat/skin interface. Under the same conditions but without the developed device, the B study group subject will have an usual behavior.

The analysis of the different behavior in these two groups will enable to evaluate, in an objective way, the potential interest of this new medical device for the prevention of pressure ulcer.

ELIGIBILITY:
Inclusion Criteria:

* patient affiliated to social security or similarly regime
* paraplegic medullary patient
* more or equal than 18 years old.

Exclusion Criteria:

patients will be excluded if at least one of the following criteria is present :

* pregnancy and feeding women
* persons without liberty by administrative or judiciary decision
* persons hospitalized without consent
* persons concerned by a justice protection action
* dependant major person
* palatine prosthesis intolerance
* buttock pressure ulcer evolution
* acute pathology (particularly mouth level)
* nickel allergy
* impossibility to use the medical device, to understand or realize the protocol due to cognitive pathologies.
* patient with dental troubles incompatible with the realisation or utilisation of orthodontic prothesis.
* no tactile feeling with tongue,
* impossibility to set up the orthodontic prothesis due to superior limb deterioration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-09; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Difference of adapted movement (in term of pressure) between the A and B groups. | 3 weeks

SECONDARY OUTCOMES:
Qualitative and quantitative knowledge evaluation | 3 weeks
Qualitative medical device evaluation | 3 weeks
Adverse event collection | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Moreau-Gaudry, Ph.D. M.D., Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital of Grenoble, Grenoble, Cedex 09, France

REFERENCES:
- [Background] Moreau-Gaudry A, Prince A, Demongeot J, Payan Y. A new health strategy to prevent pressure ulcer formation in paraplegics using computer and sensory substitution via the tongue. Stud Health Technol Inform. 2006;124:926-31. PMID 17108630